CLINICAL TRIAL: NCT00642031
Title: A Phase I Study of Triciribine Phosphate Monohydrate (TCN-PM, VD-0002) in Adult Patients With Advanced Hematologic Malignancies
Brief Title: Triciribine Phosphate Monohydrate (TCN-PM, VD-0002) in Adult Patients With Advanced Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prescient Therapeutics, Ltd. (Industry)
Collaborators: VioQuest Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0249
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Hematologic Malignancies; Leukemia
Keywords: Hematologic Malignancies; Leukemia; Chronic Myelomonocytic Leukemia; Acute Lymphocytic Leukemia; Chronic Lymphocytic Leukemia; Chronic Myelogenous Leukemia; Agnogenic Myeloid Metaplasia; Triciribine Phosphate Monohydrate; Triciribine; TCN-PM; VD-0002
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Leukemia, Myelomonocytic, Chronic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Primary Myelofibrosis | interventions — triciribine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triciribine (Experimental): Triciribine 15 mg/m^2 intravenous (IV) Weekly Over 1 Hour On Days 1, 8, and 15.
  Interventions: Drug: Triciribine

INTERVENTIONS:
Drug: Triciribine — 15 mg/m^2 IV Weekly Over 1 Hour On Days 1, 8, and 15.
  Other Names: Triciribine Phosphate Monohydrate; TCN-PM; VD-0002

SUMMARY:
Primary objective:

To determine the dose limiting toxicity (DLT) and maximum tolerated dose (MTD) of TCN-PM (Triciribine) when administered as an approximately one-hour intravenous infusion on a weekly schedule on days 1, 8 and 15 in a 28 day cycle in patients with advanced hematologic malignancies;

To determine the pharmacokinetics (PK) of Triciribine following study drug administration.

Secondary objective:

To observe the anti-tumor effects of Triciribine, if any occur

DETAILED DESCRIPTION:
Triciribine is designed to prevent development of certain proteins which participate in the abnormal growth of cancer cells.

Before you can start treatment on this study, you will have "baseline tests." These tests will help the doctor decide if you are eligible to take part in the study. You will have a physical exam, including measurement of vital signs (blood pressure, heart rate, temperature, and breathing rate). Your complete medical history will be recorded. You will be asked about your ability to perform everyday activities. You will have blood (about 4 teaspoons) and urine collected for routine tests. You will have an electrocardiogram (ECG - a test to measure the electrical activity of the heart). Women who are able to have children must have a negative blood (about 1 teaspoon) or urine pregnancy test.

You will also have a bone marrow aspiration and/or biopsy performed during the baseline testing. To collect a bone marrow aspirate and biopsy, an area of the hip or chest bone is numbed with anesthetic and a small amount of bone marrow and bone is withdrawn through a large needle.

Certain patients who are at risk for involvement of disease in their central nervous system may be required to have a lumbar puncture (spinal tap) done. A lumbar puncture involves inserting a needle between the vertebrae of the back and then removing a small amount of spinal fluid. The fluid will be checked for diseased cells, used to measure the level of study drug in the fluid, and used to measure the level of a substance that shows how the study drug is being handled by your body.

If you are found to be eligible for this study, you will start receiving Triciribine through a needle in a vein, over about 1 hour, on Days 1, 8, and 15 of each 28-day study "cycle." On each day you receive Triciribine, your vital signs will be measured before the start of the infusion, at 30 minutes (half-way through the infusion), at the end of the infusion, and at 1 hour after completing the infusion. An ECG will be done at the end of the infusion on Day 1 of the first cycle only.

The amount of Triciribine you receive in each infusion will depend on when you enter the study. At least 3 participants will be enrolled at each dose level. Each new group of participants will receive a higher dose level than the group before, unless a level is reached where the side effects are considered intolerable. This will help researchers to find out the highest tolerable dose of Triciribine.

During the study, researchers will be checking the status of the cancer to see how it is responding to the study drug. You will be checked once a week, or more often, depending on how you are doing and according to your blood cell counts. Each check-up includes measurement of your vital signs and blood (about 4 teaspoons) drawn for routine tests. You will be asked about any side effects you may have experienced and any medications you are taking.

During Cycle 1, you will have blood samples (about 1 teaspoon each time) drawn to measure the amount of study drug in your blood at different times. This is called pharmacokinetic (PK) testing. During Cycle 1, you will have a blood sample drawn before receiving the first dose of Triciribine, and then 2, 24, 48, 72 ,and 96 hours after the Day 1 Triciribine dose. If your doctor decides that it is necessary, an additional blood sample will also be drawn between 120 and 144 hours (about 5-6 days) after your Day 1 dose of Triciribine. During Cycle 1, you may also have blood samples (about 1 teaspoon) drawn to measure the action of the study drug in the tumor cells. This is called pharmacodynamic studies (this defines how the drug works on the tumor cells). During Cycle 1, you will have a blood sample drawn (about 1 teaspoon) before receiving the first dose of triciribine and then 2 and 24 hours after the Day 1 triciribine dose.

Before receiving each additional cycle, you will have a physical exam, including vital signs. Blood (about 4 teaspoons) will be drawn for routine tests, and urine will be collected. You will be asked about your ability to perform everyday activities. You will have a bone marrow exam (including aspiration and/or biopsy) about every 28 days, in order to check your response.

Certain participants who are at risk for involvement of disease in their central nervous system may be required to have repeat lumbar punctures (spinal taps) performed once a week.

You may move to a higher dose level after your first cycle of therapy, if that increased dose level is considered safe and the disease is stable or responding to treatment. If, however, you experience serious side effects from the therapy, the doctor may decide to hold any further therapy with Triciribine until those side effects go away, or may decide to stop therapy altogether, if the side effects are intolerable. Depending on how fast the side effects go away, you may be able to re-start your Triciribine infusions at a lower dose.

You may continue to receive Triciribine on study with no limit to the number of cycles that you can receive, as long as your doctor finds that you are benefiting from this therapy and you are not experiencing intolerable side effects. On the other hand, you may stop receiving the study drug and be taken off study if it is not effective for you and/or the disease gets worse, you develop another illness that interferes with the ability to safely give you the study drug, or you are unable to tolerate the study drug.

If you leave the study for any reason, you will be asked to return for a follow-up visit at the end of therapy (and possibly 30 days after your last dose of Triciribine, if you are not receiving another type of treatment). A physical exam will be performed, and blood (about 2 teaspoons) will be drawn for routine tests, during both of these visits. If you have side effects that are possibly related to the treatment, you may need to have more follow-up visits. Blood (up to 3 tablespoons) may need to be drawn for routine tests at that time.

THIS IS AN INVESTIGATIONAL STUDY. Triciribine has been authorized by the FDA for use in research only. Up to 34 patients will take part in this multicenter study. Up to 30 patients will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have relapsed/refractory leukemias for which no standard therapies are anticipated to result in a durable remission. Patients with poor-risk myelodysplasia (MDS) [i.e. refractory anemia with excess blasts (RAEB-1 or RAEB-2) by WHO classification] and chronic myelomonocytic leukemia (CMML) are also candidates for this protocol.
2. CONTINUATION # 1: Relapsed/refractory leukemias include acute non-lymphocytic leukemia (AML) by World Health Organization (WHO) classification, acute lymphocytic leukemia (ALL), chronic lymphocytic leukemia (CLL), or chronic myelogenous leukemia (CML) in blast crisis. Patients with agnogenic myeloid metaplasia (AMM) are also eligible;
3. ECOG performance status of 0- 3;
4. Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use acceptable contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device), and must have a negative serum or urine pregnancy test within 2 weeks prior to beginning treatment on this trial. Nursing patients are excluded. Sexually active men must also use acceptable contraceptive methods for the duration of time on study. Pregnant and nursing patients are excluded because the effects of Triciribine on a fetus or nursing child are unknown;
5. Must be able and willing to give written informed consent;
6. In the absence of rapidly progressing disease, the interval from prior treatment to time of study drug administration should be at least 2 weeks for cytotoxic agents, or at least 5 half-lives for noncytotoxic agents. If the patient is on hydroxyurea to control peripheral blood leukemic cell counts, the patient must be off hydroxyurea for at least 48hours before initiation of treatment on this protocol. Persistent chronic clinically significant toxicities from prior chemotherapy must not be greater than grade 1; and
7. Patients must have the following clinical laboratory values, unless abnormal parameter level is considered related to leukemia: Creatinine (Cr) less than or equal to 2.0 mg/dL, Bilirubin Normal limits (less than or equal to 1.5 * Upper Limit of Normal (ULN) with liver metastases) unless considered due to Gilbert's syndrome, Aspartate aminotransferase (AST) less than or equal to 3.0 * ULN, Alanine aminotransferase (ALT) less than or equal to 3.0 * ULN

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to uncontrolled infection, symptomatic congestive heart failure, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements;
2. Active heart disease including myocardial infarction within previous 3 months, symptomatic coronary artery disease, arrhythmias not controlled by medication, or uncontrolled congestive heart failure; and
3. Patients receiving any other standard or investigational treatment for their hematologic malignancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of TCN-PM (Triciribine) | 28 day cycle
  The MTD is the highest dose level in which <2 patients of 6 develop first cycle dose-limiting toxicity (DLT). Evaluations after each dose level (28 day cycle).

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - UT MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Sampath D, Malik A, Plunkett W, Nowak B, Williams B, Burton M, Verstovsek S, Faderl S, Garcia-Manero G, List AF, Sebti S, Kantarjian HM, Ravandi F, Lancet JE. Phase I clinical, pharmacokinetic, and pharmacodynamic study of the Akt-inhibitor triciribine phosphate monohydrate in patients with advanced hematologic malignancies. Leuk Res. 2013 Nov;37(11):1461-7. doi: 10.1016/j.leukres.2013.07.034. Epub 2013 Aug 6. PMID 23993427
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org